CLINICAL TRIAL: NCT00376090
Title: A Phase I Double-Blind, Randomized, Dose Escalating, Placebo-Controlled, Study of Safety and Immunogenicity of WRAIR/NIH Live Recombinant MVA-CMDR (HIV-1 CM235 Env/ CM240 Gag/Pol) Administered by Intramuscular (IM) or Intradermal (ID) Route In HIV-Uninfected Adults
Brief Title: Safety of and Immune Response to a Modified Vaccinia Ankara (MVA) HIV Vaccine in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RV 158; A-12403 (Other: USAMRMC HSRRB); WRAIR 1143 (Other: WRAIR HURC)
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: HIV Infections
Keywords: MVA vector; Immunogenicity; HIV vaccine; HIV preventative vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Group I Vaccine (Experimental)
  Interventions: Biological: MVA-CMDR
- Group I Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Group II Vaccine (Experimental)
  Interventions: Biological: MVA-CMDR
- Group II Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Group III Vaccine (Experimental)
  Interventions: Biological: MVA-CMDR
- Group III Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Group IV Vaccine (Experimental)
  Interventions: Biological: MVA-CMDR
- Group IV Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MVA-CMDR — 10^7 PFU IM, 1.0 mL
  Arms: Group I Vaccine
Biological: Placebo — 1.0 mL IM
  Arms: Group I Placebo; Group III Placebo
Biological: MVA-CMDR — 10^6 PFU ID, 0.1 mL
  Arms: Group II Vaccine
Biological: Placebo — 0.1 mL ID
  Arms: Group II Placebo; Group IV Placebo
Biological: MVA-CMDR — 10^8 PFU IM, 1.0 mL
  Arms: Group III Vaccine
Biological: MVA-CMDR — 10^7 PFD ID, 0.1 mL
  Arms: Group IV Vaccine

SUMMARY:
The purpose of this study is to determine the safety and the immune responses to the HIV vaccine candidate, MVA-CMDR. This vaccine was designed to induce immune responses to three HIV "passenger" genes encoded with the viral vector, MVA.

ELIGIBILITY:
Inclusion Criteria:

A participant must meet all of the following criteria:

* Low risk for HIV infection
* 18 to 40 years at the time of enrollment and vaccinia naive
* Good health
* Availability for 12 months of participation.
* Successful completion of the Test of Understanding
* Able and willing to give informed consent.
* HEMATOCRIT: WOMEN: 35 %-45 %; MEN 36 % - 49 %
* White cell count: 3,000 - 11,000 cells/mm3
* Platelets: 125,000 - 450,000 per mm3
* Normal cardiac enzyme level at second Screening Visit
* Urinalysis (UA) for protein and blood: negative or trace.
* Normal liver function tests to include ALT/AST, alkaline phosphatase, GGT (< 1.25x institutional upper limits of normal) and CPK (< 480) and creatinine (< 1.25 mg/dL)
* Negative serology for HIV infection
* Any female volunteer must have a negative serum or urine pregnancy test at the screening visit as well as immediately prior to each vaccine/placebo vaccination, as well as verbal assurance that adequate birth control measures have been followed for 60 days prior to the first vaccine/placebo vaccination and will continue to be followed for at least 3months after the final vaccine/placebo vaccination. This means using any of the following methods: Birth control drugs that prevent pregnancy given by pills, shots or placed under the skin, Male or female condoms with or without a cream or gel that kills sperm, diaphragm or cervical cap with a cream or gel that kills sperm, or Abstinence

Exclusion Criteria:

A volunteer will be excluded if one or more of the following conditions apply.

A woman who:

* Is pregnant.
* Is breast-feeding.

Anyone who:

* Is U.S. military personnel.
* Acknowledges engaging in highest-risk behavior within six months of study entry
* Has active tuberculosis or other systemic infectious process by review of systems and physical examination.
* Has history of or known cardiac disease including any of the following: prior myocardial infarction (heart attack), angina pectoris, congestive heart failure, conduction disturbances, repolarization (ST segment or T wave) abnormalities, serious cardiac arrhythmias (ventricular tachycardia or ventricular fibrillation), cardiomyopathy, pericarditis, stroke or transient ischemic attack, chest pain or shortness of breath with activity (e.g. climbing stairs), valvular heart disease including mitral valve prolapse, or other heart conditions under the care of a doctor.
* Has ECG on Screening Visit 2 with clinical significant findings, or features that would interfere with the assessment of myo/pericarditis (as determined by the contract ECG Lab) including any of the following: conduction disturbance (atrioventricular or intraventricular condition, left or right bundle branch block, AB block of any degree or QTc prolongation), repolarization (ST segment or T wave) abnormality, significant atrial or ventricular arrhythmia, frequent atrial or ventricular ectopy (e.g. frequent premature atrial contractions, 2 premature ventricular contractions in a row), ST elevation consistent with ischemia, or evidence of past or evolving myocardial infarction
* Has history of seizure disorder, immunodeficiency, chronic illness, autoimmune disease, diabetes mellitus active malignancy or use of immunosuppressive medications.
* Has evidence of psychiatric, medical and/or substance abuse problems during the past six months that the investigator believes would adversely affect the volunteer's ability to participate in the trial.
* Has occupational or other responsibilities that would prevent completion of participation in the study.
* Has received any live attenuated vaccine within 60 days of study entry.
* Has used experimental therapeutic agents within 30 days of study entry.
* Has received blood products or immunoglobulins in the past three months.
* Has history of anaphylaxis or other serious adverse reactions to vaccines.
* Has previously received an HIV vaccine or an MVA or vaccinia vaccine.
* Has chronic or active Hepatitis B or Hepatitis C virus infection or active syphilis (positive RPR and FTA).
* Has had an immediate type hypersensitivity reaction to eggs, egg products or neomycin/streptomycin (used to prepare MVA vaccine).
* Is a study site employee.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2005-07 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Study Day 0 through 8 months post-vaccination
  Evaluate the safety and tolerability of MVA-CMDR (HIV-1 CM235 Env/CM240 Gag/Pol) administered by IM or ID injection to HIV uninfected adults

SECONDARY OUTCOMES:
Immunogenicity | Study Day 0 through Study Day 280
  Evaluate the ability of MVA-CMDR (HIV-1 CM235 Env/CM240 Gag/Pol) to induce HIV antigen specific cellular and humoral immune responses

CONTACTS AND LOCATIONS:
Overall Officials: Mary Marovich, MD, DTM&H, Principal Investigator — US Military HIV Research Program
Locations (1):
- US Military HIV Research Program, Rockville, Maryland, United States

REFERENCES:
- [Derived] Currier JR, Ngauy V, de Souza MS, Ratto-Kim S, Cox JH, Polonis VR, Earl P, Moss B, Peel S, Slike B, Sriplienchan S, Thongcharoen P, Paris RM, Robb ML, Kim J, Michael NL, Marovich MA. Phase I safety and immunogenicity evaluation of MVA-CMDR, a multigenic, recombinant modified vaccinia Ankara-HIV-1 vaccine candidate. PLoS One. 2010 Nov 15;5(11):e13983. doi: 10.1371/journal.pone.0013983. PMID 21085591